CLINICAL TRIAL: NCT02505087
Title: Pharmacological Treatment of a Rare Genetic Disease: Pilot Trial Phase II-III With N-acetylcysteine in Myopathy Associated SEPN1-RM (Selenoprotein N-related Myopathy)
Brief Title: Pharmacological Treatment of a Rare Genetic Disease: N-acetylcysteine in Myopathy Associated Selenoprotein N-related Myopathy (SEPN1-RM)
Acronym: SelNac
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P100152
Record Dates: First submitted 2015-06-25; First posted 2015-07-22 (Estimated); Last update posted 2020-09-29 (Actual); Status verified 2017-11

CONDITIONS: Selenoprotein N-related Myopathy
Keywords: Selenoprotein N-related myopathy; biomarkers; washout; N-ACETYLCYSTEINE

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo followed by N-Acetylcysteine (Active Comparator): Arm receiving placebo for 6 months, then N-Acetylcysteine (NAC) for 6 months.
  Interventions: Drug: Placebo followed by N-Acetylcysteine
- N-Acetylcysteine followed by Placebo (Experimental): Arm receiving N-Acetylcysteine (NAC) for 6 months and then placebo for 6 months.
  Interventions: Drug: N-Acetylcysteine followed by Placebo
- Healthy volunteers (No Intervention): The purpose of this group is to collect reference values for biochemical markers.

INTERVENTIONS:
Drug: N-Acetylcysteine followed by Placebo — Arm receiving N-Acetylcysteine (NAC) for 6 months and then placebo for 6 months.
  Treatment periods are separated by a 2 month washout.
  Arms: N-Acetylcysteine followed by Placebo
Drug: Placebo followed by N-Acetylcysteine — Arm receiving placebo for 6 months then N-acetylcysteine (NAC) for 6 months. Treatment periods are separated by a 2 month washout.
  Arms: Placebo followed by N-Acetylcysteine

SUMMARY:
The objective of this study is to determine whether the administration of N-acetylcysteine (NAC) improves oxidative stress. To determine this, the study will assess the impact of oral treatment on the balance between reduced and oxidized form of glutathione in erythrocytes of peripheral blood.

DETAILED DESCRIPTION:
A prospective, monocentric, crossover, double-blind, placebo-controlled study.

For each patient the study will be divided in two treatment periods of 6 months separated by a 2 month washout period. 24 patients will be randomized in two groups, one group treated first with placebo during 6 months, followed by 6 months; the second group treated in the reverse sequence, then placebo.

24 healthy volunteers will also be enrolled in the study in order to collect reference values for biochemical biomarkers.

D-1: run-up visit, patients will be hospitalized in intensive care unit to collect information about diet, physical activity and smoking.

During follow-up visits: we will analyze the impact of treatment with N-acetylcysteine (NAC) on:

* Biomarkers of redox homeostasis,
* Measures of locomotor functional capacity,
* Body mass composition,
* Respiratory functional abilities.

Biomarkers that reflect the status of antioxidant defense mechanisms, parameters that reflect the cell damage to oxidative stress, the markers of inflammation and metabolic alterations induced by oxidative stress, body composition in terms of lean mass and fat mass, the motor functional abilities, respiratory function capabilities, will be compare before and after treatment.

These measures could complement the information on the status of oxidative stress and clarify the effects of N-acetylcysteine (NAC) on the evolution of the disease in these patients.

The correlation of biomarker measurements in muscle and systemic tissues will be checked.

Furthermore we will collect information about the lifestyle through standardized questionnaires that include diet, smoking, and habitual physical activity. Environmental factors and lifestyle can influence the balance oxidant / antioxidant patients and contribute to the variability of the clinical severity of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. For patients:

   * Patient >18 and <60 years old
   * Patients with Selenoprotein N-related myopathy with homozygous or compound heterozygous mutations in the gene SEPN1-RM
   * Informed written consent
   * Patients capable of being followed up throughout the duration of the study
   * Patient trained in the use of cough assist
   * Patients having an health insurance
   * Patient accepting to commit not to introduce major changes in diet and lifestyle during the study period
2. For healthy volunteers:

   * volunteers >18 and <60 years old
   * Informed written consent
   * Health insurance

Exclusion Criteria:

1. For patients:

   * Pregnancy
   * Intolerance to N-acetylcysteine (NAC), galactose or fructose; malabsorption glucose or galactose; lactase deficiency
   * Consumption of synthetic vitamins, NAC and other antioxidants within 3 months prior to inclusion
   * Treatment with corticosteroids or non-steroidal anti-inflammatory from time to time in the 4 weeks preceding the inclusion or for more than 3 days between 12 and 4 weeks before inclusion
   * Planned surgery within 3 months before inclusion or during the inclusion period
   * Intercurrent or existing illnesses such as chronic infectious diseases (HIV, hepatitis, etc.), asthma, malignant tumor pathology, Hematological Pathology
   * Expected survival less than 14 months
   * Inability to understand the instructions or the implications of the Protocol
2. For healthy volunteers:

   * Pregnancy
   * Consumption of synthetic vitamins, NAC and other antioxidants within 3 months prior to inclusion
   * Treatment with corticosteroids or non-steroidal anti-inflammatory from time to time in the 4 weeks preceding the inclusion or for more than 3 days between 12 and 4 weeks before inclusion
   * Planned surgery within 3 months before inclusion or during the inclusion period
   * Intercurrent or existing illnesses such as chronic infectious diseases (HIV, hepatitis, etc.), asthma, malignant tumor pathology, Hematological Pathology
   * Inability to understand the instructions or the implications of the Protocol
   * Bleeding disorders or other bleeding risks or risk of infection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Ratio of reduced glutathione and oxidized glutathione in blood erythrocytes. | 6 months in each period

SECONDARY OUTCOMES:
measure of health status according The 36-Item Short Form Health Survey (SF36) | 6 months in each crossover period
Evaluate the impact of fatigue according the Fatigue Severity Scale (FSS) | 6 months in each crossover period
Measurement of biomarkers in blood samples, muscle and fibroblasts | 6 months in each crossover period
Measure of Activity Limitation (Activlim test) | 6 months in each crossover period
Running speed measured by the test of 10 m | 6 months in each crossover period
Measures of motor function according a Motor Function Measure scale (MFM ) | 6 months in each crossover period
Muscular endurance is measured by the test of 2 minutes walk | 6 months in each crossover period
Measurement of the maximum voluntary contraction of the quadriceps | 6 months in each crossover period
The measurement of the endurance of the quadriceps | 6 months in each crossover period
Assessment of dyspnea according Borg scale | 6 months in each crossover period

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte ESTOURNET, MD, PhD, Principal Investigator — Neuro-Respiratory Rehabilitation Service, Raymond Poincaré Hospital, 92380 Garches, France
Locations (1):
- UMR8251 University Paris Diderot / CNRS, Paris, France